CLINICAL TRIAL: NCT01946984
Title: Intramuscular Diclofenac vs. Placebo in a Randomized Double Blind Controlled Trial, In Post ERCP Pancreatitis.
Brief Title: Diclofenac vs. Placebo in a Randomized Double Blind Controlled Trial in Post ERCP Pancreatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Specialized Arab Hospital (Other)
Responsible Party: Principal Investigator, Yasser Abu-Safieh, Associate Prof, MD, AGAF, Specialized Arab Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Specialized Arab Hospital
Record Dates: First submitted 2013-09-09; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Post-ERCP Acute Pancreatitis.
Keywords: diclofenac, ERCP and pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Cholangiopancreatography, Endoscopic Retrograde; diclofenac hydroxyethylpyrrolidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diclofenac,75 mg, 3 ml, (Active Comparator): patients were given Diclofenac IM before ERCP.
  Interventions: Procedure: ERCP; Drug: Diclofenac hydroxyethylpyrrolidine
- Normal Saline, 3ml, IM (Placebo Comparator): patients were given normal saline 3 ml before ERCP
  Interventions: Procedure: ERCP; Drug: Normal Saline

INTERVENTIONS:
Procedure: ERCP — endoscopy, retrograde cholangio-pancreaticography.
Drug: Diclofenac hydroxyethylpyrrolidine
  Arms: Diclofenac,75 mg, 3 ml,
Drug: Normal Saline
  Arms: Normal Saline, 3ml, IM

SUMMARY:
1. The most common complication of endoscopic retrograde cholangio-pancreaticography (ERCP) is pancreatitis.
2. Several studies showed that non-steroidal anti-inflammatory drugs (NSAIDs) can prevent the post ERCP pancreatitis, the investigators used diclofenac vs placebo.
3. The effect of diclofenac in prevention of that complication, was measured by the number of patients who developed pancreatitis, and compare it with the placebo.
4. The investigators collected 199 patients, 17 excluded, 182 completed the study, all of them underwent the intervention called "ERCP", and randomized to have either Diclofenac or Placebo before the procedure.

DETAILED DESCRIPTION:
* All patients signed informed consents for the procedure, and the participation in the study.
* Between June 2012 and June 2013, 199 patients fulfilled the inclusion criteria, 182 of whom were included in the final analysis.
* Patients were excluded from study participation if they had a contraindication for diclofenac, including patients with recently diagnosed peptic ulcer disease, renal failure, those who developed acute pancreatitis during the two weeks before ERCP, those with a history of chronic pancreatitis, and those who did not agree to participate in the study.
* A placebo-controlled trial was conducted in 182 patients who underwent ERCP.
* Preoperative, the patients received 75 mg intramuscular(IM) diclofenac or IM normal saline as placebo. At the end of each procedure, the investigators recorded the details of the maneuvers performed, including:

  1. the total time of the procedure,
  2. the number of attempts at cannulation,
  3. the number of pancreatic duct cannulation,
  4. the final diagnosis by ERCP,
  5. whether a sphincterotomy, a needle-knife papillotomy, or stent placement were performed.
* Serum amylase was determined 12 hours after ERCP.

  * If the 12-hours serum amylase level was > 3 times the upper normal limit and the patient exhibited pain or nausea and vomiting, then the patient had pancreatitis.
  * Acute pancreatitis was defined as serum amylase > 3 times the upper limit of normal and associated with epigastric pain, back pain, and epigastric tenderness.
* Statistical analysis:

  1. Randomization was done by the GI nurse, concealed envelop
  2. Data were summarized by descriptive statistics.
  3. The Chi square was used to compare categorical patient data.
  4. The Student's t test was used to compare continuous variables.
  5. Two-tailed P < 0.05 was considered to indicate significance.

ELIGIBILITY:
Inclusion Criteria:

* any patient above the age of 16, referred for ERCP

Exclusion Criteria:

* 1.could not reach the ampulla due to: A. Pyloric stenosis B. Ampullary tumor C. Diverticula 2. ERCP done recently 3. Stent replacement 4. Congestive Heart Failure(CHF) 5. Asthma

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
prevention of pancreatitis, | within a week after procedure
  1. Patients with epigastric pain, back pain, and epigastric tenderness,
  2. And all had serum amylase measured after the procedure, if elevated more than 3 folds of normal, the patient was diagnosed to have post ERCP pancreatitis,

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Abu-Safieh, MD, AGAF, Principal Investigator — Specialized Arab Hospital
Locations (1):
- SAH hospital, Nablus, West Bank, Palestinian Territories